CLINICAL TRIAL: NCT03513536
Title: The Effect of Scent on Pregnancy Induced Nausea, Vomiting, and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-2300
Record Dates: First submitted 2018-04-05; First posted 2018-05-01 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Morning Sickness; Pregnancy Early
Keywords: Aromatherapy; Essential Oils
MeSH Terms: conditions — Morning Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention 1 (Experimental): The women in this arm will receive the Citrus-Based Aromatherapy product to apply regularly for 6 days.
  Interventions: Other: Citrus-Based Aromatherapy
- Intervention 2 (Experimental): The women in this arm will receive the Mint-Based Aromatherapy product to apply regularly for 6 days.
  Interventions: Other: Mint-Based Aromatherapy
- Intervention 3 (Experimental): The women in this arm will receive the Spice-Scented Aromatherapy product to apply regularly for 6 days.
  Interventions: Other: Spice-Scented Aromatherapy
- Control (Placebo Comparator): The women in this arm will receive a vegetable oil roll-on product to apply regularly for 6 days.
  Interventions: Other: Control

INTERVENTIONS:
Other: Citrus-Based Aromatherapy — This intervention is a blend of plant derived oils which have been distilled from crude plant matter and analyzed in a laboratory to identify chemical composition.
  Arms: Intervention 1
Other: Mint-Based Aromatherapy — This intervention is a blend of plant derived oils which have been distilled from crude plant matter and analyzed in a laboratory to identify chemical composition.
  Arms: Intervention 2
Other: Spice-Scented Aromatherapy — This intervention is a blend of plant derived oils which have been distilled from crude plant matter and analyzed in a laboratory to identify chemical composition.
  Arms: Intervention 3
Other: Control — This control is a blend of plant derived oils which have been expressed from crude plant matter.
  Arms: Control

SUMMARY:
This study evaluates the effects of essential oils on nausea, vomiting, and quality of life scores among pregnant women. Participants will receive either an essential oil roll-on product or a placebo product to apply to their temples and jaw line daily for 6 days.

DETAILED DESCRIPTION:
The inhalation of certain essential oils has been found to reduce feelings of nausea and to improve quality of life during pregnancy.

The essential oils used in this study are applied topically to the temples and jaw line every 4-6 waking hours over a 6-day period. Each application will produce an exposure that lasts up to 30-45 minutes before fading. At the end of each day, nausea and vomiting levels will be assessed using a validated measurement instrument.

Quality of life is measured using a 30-question tool that measures both pregnancy-related quality of life and pregnancy-induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-45 years
* confirmed pregnancy
* healthy pregnancy

Exclusion Criteria:

* hyperemesis gravidarum
* tobacco use in the home
* high risk pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Change from Nausea and Vomiting 6-part Quantification of Emesis scale | daily for 6 days
  Nausea and vomiting are measured once per day using the 6-item Quantification of Emesis 24-hour scale (PUQE) scale. This scale includes 3 questions which are ranked on a scale of 1-5, with higher scores indicating higher levels of pregnancy-induced nausea and vomiting. The other 3 questions are open-ended questions which ask participants about perceived well-being.

SECONDARY OUTCOMES:
Health Related Quality of Life for Nausea and Vomiting of Pregnancy 30-part scale | baseline and day 6
  Quality of life is measured twice, at the start of the study and at the end of the study, using the Health Related Quality of Life for Nausea and Vomiting of Pregnancy (NVPQOL) instrument. This instrument includes 30 questions which are ranked on a Likert scale with 1 indicating "none of the time" and 7 indicating "all of the time." Higher scores indicate higher levels of nausea and vomiting, with reduced quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Hawkins, PhD, Principal Investigator — Nutraceuticals Research Institute
Locations (1):
- Franklin Institute of Wellness, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share